CLINICAL TRIAL: NCT02962765
Title: Prospective, Multinational, Non-interventional Post-authorisation Study to Document the Long-term Immunogenicity, Safety, and Efficacy of Human-cl rhFVIII (Simoctocog Alfa) in Patients With Haemophilia A Treated in Routine Clinical Practice
Brief Title: Non-interventional Post-authorisation Study to Document the Immunogenicity, Safety, and Efficacy of NUWIQ
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GENA-99
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Citrate Plasma for measuring FVIII inhibitors is recommended throughout the study.
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, multinational, non-interventional post-authorisation study to collect additional clinical data and to ensure consistency in the long-term between the outcome from pre-authorisation clinical studies (in 135 previously treated paediatric and adult patients) and routine clinical practice. Besides aspects such as general product safety and efficacy, there will be a focus on immunogenicity, particularly on inhibitor development. The diagnosis of FVIII inhibitor will be based on clinical observations and confirmed by FVIII inhibitor testing in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A (FVIII:C ≤ 2%) based on medical history; at least 100 patients should have severe haemophilia A (FVIII:C < 1%)
* Male patients of any age
* Previous treatment with a FVIII concentrate for more than 150 EDs
* Availability of detailed documentation (patient diary, log book, etc.) covering either the last 50 EDs or the last 2 years per patient to confirm treatment modality (i.e., prophylaxis, on-demand, recent surgery, or immune tolerance induction)
* Inhibitor negative (< 0.6 BU) at study entry as confirmed by a recovery test with previous FVIII product and inhibitor test in a central laboratory
* Immunocompetence (CD4+ count > 200/µL), HIV-negative, or having a viral load < 200 particles/µL or < 400,000 copies/mL
* Decision to prescribe Human-cl rhFVIII before enrolment into the study
* Written informed consent by the patient or the patient's parent or legal guardian

Exclusion Criteria:

* Patients treated with any investigational medicinal product (IMP) except FVIII IMP within 30 days prior to the Screening Visit or patients planning to undergo treatment with any IMP other than Human-cl rhFVIII are not eligible for enrolment into the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The goal is to collect data on 200 previously treated male patients of any age with haemophilia (FVIII:C ≤ 2%). Patients from pre-authorisation studies can be followed up to at least 100 EDs. Newly enrolled patients have to be treated and followed for at least 100 EDs.
  * Of the 200 enrolled patients, at least 100 patients should have severe haemophilia A (FVIII:C < 1%).
  * Of the 200 enrolled patients, approx. 60 patients should be < 12 years of age. At least 10 patients should be aged between 14-18 years.
  * Patients with severe haemophilia A after successful immune tolerance induction (ITI) can also be included; the proportion of these ITI patients should not exceed 25% of the entire cohort.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Khair, PhD, Principal Investigator — Great Ormond Street Hospital
Locations (39):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Tulane University, New Orleans, Louisiana
  - Hemophilia Treatment Center of Nevada, Las Vegas, Nevada
  - Gulf States Hemophilia and Thrombophilia, Houston, Texas
- Argentina (4):
  - Centro de Tratamiento de la Hemofilia Cordoba, Córdoba
  - CTH Centro de Tratamiento de Hematologia y Hemoterapia Córdoba S.A., Córdoba
  - Fundación de Hemofilia de Salta, Salta
  - Centro Mayo, Santiago del Estero
- Belarusian Research Center for Pediatric Oncology, Hematology and Immunology, Borovlyany, Belarus
- Czechia (2):
  - Fakultní nemocnice Brno, Brno
  - Blood Centre, University Hospital, Ostrava
- Hospital de Especialidades Teodoro Maldonado Carbo, Guayaquil, Ecuador
- France (4):
  - CHU Hôtel Dieu, Nantes
  - Hopital Pontchaillou, Rennes
  - CHRU Hôpital Nord, Saint-Priest-en-Jarez
  - CRTH, Hopital Purpan, Toulouse
- Pedias Inc. Centro Hospitalario La Paz, Guatemala City, Guatemala
- Italy (13):
  - L'Azienda Ospedaliero Universitaria Consorziale Policlinico, U.O. di Medicina Trasfusionale, Centro Emofilia e Trombosi, Bari
  - U.O.C. Ematologia, Ospedale San Giacomo Apostolo, Castelfranco Veneto
  - UOC Malattie emorragiche e della coagulazione, Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Ca Granda, Milan
  - AOU Federico II - Dipartimento di Medicina Clinica e Chirurgica, Naples
  - Azienda Sanitaria Locale Napoli 1 Centro, Naples
  - Azienda Ospedaliera di Padova, Padua
  - AOU Policlinico di Palermo, Palermo
  - Ospedale ARNAS Civico, Palermo
  - Dipartimento Di Medicina dell'Universita degli Studi di Perugia, Perugia
  - Dipartimento di Biotecnologie Cellulari ed Ematologia -"Sapienza" Università di Roma, Rome
  - A.O. Città della Salute e della Scienza di Torino - Ospedale Regina Margherita, Torino
  - S.C. Ematologia U, A.O.U. Città della Salute e della Scienza di Torino, Torino
- Vilnius University Hospital, Santariskiu Klinikos-Children's Hospital, Vilnius, Lithuania
- Oslo University Hospital, Oslo, Norway
- Centro Hospitalar Cova da Beira, Covilha, Portugal
- National Haemophilia Center, Bratislava, Slovakia
- United Kingdom (4):
  - Great Ormond Street Hospital (GOSH), London
  - St. Thomas' Hospital, London
  - The Royal London Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

RESULTS

PARTICIPANT FLOW:
Groups:
- Nuwiq® (Human-cl rhFVIII): A total of 80 patients were enrolled in this study.
  Of the 80 patients enrolled into the study, 2 were excluded because they had not received any treatment with Nuwiq, leaving 78 patients in the full analysis population (FAS) and safety population (SAF).
  Of these, 77 patients were part of the prophylactic treatment group and 2 patients were in the on-demand treatment group.
  One patient changed regimen from on-demand treatment to prophylactic treatment and back to on-demand treatment while in the study. Corresponding data for this patient in included in both the prophylactic and on-demand treatment groups.
  The treatment regimen, doses, dosing intervals and dose adjustments were determined at the discretion of the treating physician. A usual dose for long-term prophylaxis against bleeding in patients with severe hemophilia A is 20 to 40 IU of factor VIII per kg body weight at intervals of 2 to 3 days.
  Of the 78 total patients, 17 were excluded for the reasons summarized below.
Period: Overall Study
Arm/Group | Nuwiq® (Human-cl rhFVIII)
Started | 78
FAS Population | 78
SAF Population | 78
Prophylactic Treatment Group | 77
On Demand Treatment Group | 2
SURG Population | 4
Completed | 61
Not Completed | 17
Not completed — Protocol Violation | 9
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Limited access to study medication | 3

BASELINE CHARACTERISTICS:
Groups:
- Nuwiq® (Human-cl rhFVIII) SAF Population: The safety (SAF) population consist of all patients who received at least one infusion of Human-cl rhFVIII (n=78)
Arm/Group | Nuwiq® (Human-cl rhFVIII) SAF Population
Number analyzed (Participants) | 78
Age, Customized [Count of Participants; unit: Participants]
  Age: <12 yrs | 40
  Age: 12-<18 yrs | 12
  Age: >18 yrs | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Patient race: American Indian or Alaska Native | 7
  Patient race: Asian | 0
  Patient race: Native Hawaiian or Other Pacific Islander | 0
  Patient race: Black or African American | 1
  Patient race: White | 61
  Patient race: More than one race | 0
  Patient race: Other | 9
Height [Mean (Standard Deviation); unit: centimeters]
  <12 yrs | 112 (17.59)
  12-<18 yrs | 168.8 (9.73)
  >18 yrs | 172.9 (7.88)
Weight [Mean (Standard Deviation); unit: kilograms]
  <12 yrs | 21.7 (8.30)
  12-<18 yrs | 67.1 (15.55)
  >18 yrs | 76.6 (17.21)
BMI [Mean (Standard Deviation); unit: kg/m^2]
  <12 yrs | 17.0 (3.34)
  12-<18 yrs | 23.6 (5.46)
  >18 yrs | 25.5 (4.65)
Severity of Haemophilia A [Count of Participants; unit: Participants] — Moderate Hemophilia was defined as the patient having a FVIII activity level of between 1-2%. Severe Hemophilia was defined as the patient having a FVIII activity level below 1%.
  Participants
    Moderate | 10
    Severe | 68
Family history of Haemophilia [Count of Participants; unit: Participants]
  Yes | 47
  No | 31
Factor VIII Inhibitor History [Count of Participants; unit: Participants]
  Yes | 10
  No | 68
Factor VIII gene defect [Count of Participants; unit: Participants]
  Intron 22-Inversion | 17
  Large Deletion/Insertion | 1
  Small Deletion/Insertion | 5
  Stop-Mutation | 4
  Nonsense Mutation | 4
  Missense Mutation | 2
  Other | 9
  Unknown | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With FVIII Inhibitors
Description: FVIII inhibitors will be determined based on clinical observations and confirmed by FVIII inhibitor testing in the laboratory.
Time Frame: Screening through to study completion (minimum 1.7 months; maximum 31.6 months)
Population: FVIII inhibitor testing could be carried out at any time at the physician's discretion. Patients were checked for clinical symptoms suggesting FVIII inhibitor development, any suspicion of inhibitor formation was to be investigated by FVIII inhibitor testing. No symptoms led to suspicion of inhibitor formation in any patient treated with Nuwiq®. Within the FAS population, inhibitor levels were tested in 40 patients at screening, 44 between screening and completion and 21 at study completion.
Measure: Count of Participants; unit: Participants
Groups:
- FVIII Inhibitors Detected at Screening in Patients Treated With Nuwiq®: FVIII inhibitors detected in the FAS population at screening.
- FVIII Inhibitors Detected Between Screening and Completion in Patients Treated With Nuwiq®: FVIII inhibitors detected in the FAS population between screening and study completion
- FVIII Inhibitors Detected at Completion in Patients Treated With Nuwiq® (Human-cl rhFVIII): FVIII inhibitors detected in the FAS population at study completion
Arm/Group | FVIII Inhibitors Detected at Screening in Patients Treated With Nuwiq® | FVIII Inhibitors Detected Between Screening and Completion in Patients Treated With Nuwiq® | FVIII Inhibitors Detected at Completion in Patients Treated With Nuwiq® (Human-cl rhFVIII)
Number analyzed (Participants) | 40 | 44 | 21
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Adverse Drug Reactions
Description: Adverse drug reactions (ADRs) including hypersensitivity reactions will be recorded by patients in treatment diaries which will be reviewed at each Follow-up Visit.
Time Frame: Recorded from screening through to study completion (minimum 1.7 months; maximum 31.6 months)
Measure: Count of Participants; unit: Participants
Groups:
- Nuwiq® (Human-cl rhFVIII) FAS Population: All patients who received at least one infusion of Nuwiq® (Human-cl rhFVIII) and for whom at least one measurement after screening was available
Arm/Group | Nuwiq® (Human-cl rhFVIII) FAS Population
Number analyzed (Participants) | 78
Participants | 0

3. Secondary Outcome: Annualized Rate of Breakthrough Bleeds to Assess Efficacy in Prophylactic Treatment
Description: Total number of bleeding episodes under prophylaxis treatment divided by the duration of prophylactic phase (in years)
Time Frame: Monitored throughout the study from screening through to study completion (minimum 3.7 months; maximum 21.2 months)
Population: Of the 77 participants within the prophylactic treatment group, 74 patients had at least 3 months under a prophylactic regimen and had at least one bleeding episode and were analyzed.
Measure: Median (Inter-Quartile Range); unit: Number of bleeding episodes per year
Units Other Than Participants: Number of bleeding episodes
Groups:
- Nuwiq® in Prophylactic Treatment: Patients with at least 3 months routine prophylactic treatment with Nuwiq
Arm/Group | Nuwiq® in Prophylactic Treatment
Number analyzed (Participants) | 74
Number analyzed (Number of bleeding episodes) | 252
Number of bleeding episodes per year
  All bleeding events | 2.39 [0 to 4.87]
  Spontaneous bleeding events | 0.00 [0 to 2.47]
  Traumatic bleeding events | 0.00 [0 to 1.93]

4. Secondary Outcome: Assessment of the Efficacy of On-demand Treatment of Bleeding Episodes (BEs) Based on a 4-point Efficacy Scale
Description: At the end of a BE, treatment efficacy was to be assessed either by the patient (or the patient's parent or legal guardian) or by the treating physician in case of on-site treatment using a 4-point scale including the four items 'excellent,' 'good,' moderate,' and 'none.' Excellent result was defined as abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single injection. Good was definite pain relief and/or improvement in signs of bleeding within approximately 8-12 hours after an injection requiring up to 2 injections for complete resolution. Moderate was probable or slight beneficial effect within approximately 12 hours after the first injection requiring more than two injections for complete resolution. None was no improvement after 12 hours, or worsening of symptoms, requiring more than 2 injections for complete resolution.
Time Frame: Monitored throughout the study from screening through to study completion (minimum 1.7 months; maximum 31.6 months)
Measure: Number; unit: Number of Bleeding episodes
Units Other Than Participants: Number of bleeding episodes
Groups:
- Nuwiq® (Human-cl rhFVIII) in On Demand Population: Efficacy of Nuwiq in the treatment of bleeding episodes (BEs) in patients who were under on-demand treatment
Arm/Group | Nuwiq® (Human-cl rhFVIII) in On Demand Population
Number analyzed (Participants) | 2
Number analyzed (Number of bleeding episodes) | 55
Number of Bleeding episodes
  Excellent | 50
  Good | 4
  Moderate | 1
  None | 0

5. Secondary Outcome: Overall Assessment of the Effectiveness of Surgical Prophylaxis by the Treating Physicians
Description: At the end of the postoperative period, an overall assessment of the efficacy of treatment in the pre-, peri-, and postoperative periods using the 'excellent,' 'good,' moderate,' and 'none' scale will be done jointly by the surgeon and the hematologist. Based on this assessment, efficacy ratings assessed as either 'excellent' or 'good' will be considered 'successfully treated'.
Time Frame: From start of surgery until end of post-operative period
Population: A total of 4 patients had 6 surgeries that were treated with Nuwiq®. Two of these surgeries were minor and 4 were major. Five surgeries had an overall efficacy assessment performed jointly by the hematologist and surgeon. One of the six surgeries was treated pre-op with another FVIII product and post-op with Nuwiq® and therefore an assessment of Nuwiq® efficacy could not be performed
Measure: Number; unit: Surgeries
Units Other Than Participants: Surgeries
Groups:
- Nuwiq® (Human-cl rhFVIII) Surgical Prophylaxis: 4 patients had in total 6 surgeries and were included in the SURG population.
Arm/Group | Nuwiq® (Human-cl rhFVIII) Surgical Prophylaxis
Number analyzed (Participants) | 4
Number analyzed (Surgeries) | 5
Surgeries
  Excellent | 5
  Good | 0
  Moderate | 0
  None | 0

6. Secondary Outcome: Assessment of the Efficacy of Treatment of Bleeding Episodes (BEs) Based on a 4-point Efficacy Scale
Description: At the end of a BE, treatment efficacy was to be assessed either by the patient (or the patient's parent or legal guardian) or by the treating physician in case of on-site treatment using a 4-point scale including the four items 'excellent', 'good', 'moderate', and 'none.'
  Excellent result was defined as abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single injection. Good was definite pain relief and/or improvement in signs of bleeding within approximately 8-12 hours after an injection requiring up to 2 injections for complete resolution. Moderate was probable or slight beneficial effect within approximately 12 hours after the first injection requiring more than two injections for complete resolution. None was no improvement after 12 hours, or worsening of symptoms, requiring more than 2 injections for complete resolution.
Time Frame: Recorded from screening through to study completion (minimum 1.7 months; maximum 31.6 months)
Population: Analysis was only performed on patients in the prophylactic treatment group who experienced bleeding episode that required treatment with Nuwiq. Of the 77 patients in the prophylactic treatment group, 48 patients experienced a BE that required treatment with Nuwiq and were assessed using the 4-point efficacy scale
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Number of treated Bleeding episodes
Groups:
- Nuwiq in Prophylactic Population: Efficacy of Nuwiq in the treatment of bleeding episodes in patients who were under prophylactic treatment
Arm/Group | Nuwiq in Prophylactic Population
Number analyzed (Participants) | 48
Number analyzed (Number of treated Bleeding episodes) | 246
Bleeding episodes
  Excellent | 167
  Good | 50
  Moderate | 26
  None | 3

ADVERSE EVENTS:
Time Frame: Adverse drug reactions were monitored throughout the study from first treatment through to study completion (minimum 1.7 months; maximum 31.6 months)
Description: One death was recorded during the study. The patient was reported as having died due to a possible intentional/unintentional overdose of prescribed medications (not Nuwiq®). The investigator reported no suspected relationship between Nuwiq® and the death of the patient and the event was deemed unrelated to Nuwiq®.
Groups:
- Nuwiq® (Human-cl rhFVIII) SAF Population: Adverse events were reported for the SAF population which consist of all patients who received at least one infusion of Human-cl rhFVIII (n=78). Due to no reported adverse events related to treatment with Nuwiq, AEs were not reported separately for prophylactic or on-demand interventions.
Arm/Group | Nuwiq® (Human-cl rhFVIII) SAF Population
All-Cause Mortality (participants affected / at risk) | 1/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02962765/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02962765/SAP_001.pdf